CLINICAL TRIAL: NCT06753344
Title: Youth Promotion of Resilience Involving Mental E-health
Acronym: Y-PRIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: St. Francis Xavier University (Unknown); Institute of Population, Health and Development, Vietnam (Other); Simon Fraser University (Other); University of Melbourne (Other)
Responsible Party: Principal Investigator, Raymond Lam, MD, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H24-01700
Record Dates: First submitted 2024-12-17; First posted 2024-12-31 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Mental Well-being; Resilience; Population Study
Keywords: digital mental health; youth; LMIC; well-being; resilience; life skills education
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The experimental arm will use our app-based intervention [name TBD] at their own pace for 1 year. The app will introduce and teach six life and self-management skills to promote general mental well-being and resilience among Vietnamese youth. During the year, they will complete the outcome survey at baseline, 6 months, and 12 months marks. App data will be collected.
  Interventions: Behavioral: Intervention app
- Control group (No Intervention): The no intervention arm will complete the outcome survey at baseline, 6 months, and 12 months. After 12 months, they will gain access to the intervention app (at the same time as the experimental group) but no app data will be collected.

INTERVENTIONS:
Behavioral: Intervention app — The app-based intervention, co-designed with the V-YAC, aims to introduce life skills and self-management skills to promote general mental well-being and resilience among Vietnamese youth. With this app, youth users will have a fun and safe space to learn and practice six life skills areas (Problem-solving, Social Media and Well-being, Communication and Interpersonal Skills, Realistic Thinking, Coping with Emotions and Stress, and Goal Setting). Lessons (in the form of short texts) and activities (ex. multiple choice activities, blank worksheets, reflection questions) were adapted from evidence-based interventions developed in other contexts to be culturally appropriate to the Vietnamese youth context. Youth users are free to explore the app at their own pace. Gamification features will also allow youth users to collect points in the app for completing each lesson, activity, or challenge.
  Arms: Intervention Group

SUMMARY:
There is a critical gap in access to mental health promotion, prevention and support among youth worldwide, especially in low and middle-income countries like Vietnam. The Y-PRIME Study aims to respond to this gap by co-designing with Vietnamese youth a mobile app that delivers life skills and self-management skills intervention to promote mental well-being in grade 10 Vietnamese students. Working with the Vietnam Youth Advisory Council (V-YAC) to adapt and co-design the intervention and app ensure that the intervention will be culturally appropriate and relevant to Vietnamese youth. The goal of the current phase is to test this intervention with grade 10 students across three provinces (Hanoi, Thai Binh, and Hung Yen) to assess:

1. Whether the app helps to improve mental well-being and resilience among youth in Vietnam and helps to reduce factors that might increase the risk of poor mental well-being, like stress related to school and other pressures
2. Whether the app can be delivered in Vietnamese schools
3. Whether Vietnamese youth and school staff think the app is appropriate and appealing for youth in order to scale-up the model across the country

The control group (meaning they do not have access to the app-based intervention) will complete the outcome survey at baseline, 6 months, and 12 months. After 12 months, they will gain access to the intervention app (at the same time as the experimental group) but no more data will be collected. The intervention group will use the app at their own pace for 1 year while completing the same survey at baseline, 6 months, and 12 months marks. Afterwards, students and school health staff will be invited to a focus group discussion to talk about their experience using the app.

DETAILED DESCRIPTION:
Between 10-20% of the world's children and youth experience mental health problems; suicide is among the five leading causes of mortality among adolescents. Despite this, youth-oriented mental health promotion, prevention, and support are severely limited, especially in low and middle-income countries (LMICs). Vietnam has a population of 97 million people, 70% of whom are under the age of 35 years. Like many LMICs, Vietnam has extremely limited mental health promotion, prevention and care availability for youth. Life skills-based programs, delivered at a population level via schools, are an evidence-based approach that have the potential to improve mental health, resilience, and well-being among youth in low- resource settings. Digital health approaches including interventions delivered via mobile apps are also increasingly recognized as an effective, acceptable, and accessible approach to promoting youth mental health and wellness and warrant more research, particularly within LMICs.

The Youth Promotion of Resilience Involving Mental E-health (Y-PRIME) study will respond to the gap in the availability of evidence-based interventions to promote mental health, well-being, and resilience for youth in Vietnam. In Phase 1 of the study, the investigators engaged key stakeholders in the adaptation and co-design of an evidence-based mobile app intervention to be used among secondary school students. In this current study, the mobile app will be tested among secondary school students in three provinces (Hanoi, Thai Binh, Hung Yen) in Vietnam.

The investigators hypothesize that a youth-informed intervention adapted for the Vietnamese context and delivered via an app will lead to positive implementation outcomes among youth and within the implementation environment. The investigators also posit that it will lead to improved mental health, well-being, resilience, and risk-factor-related outcomes among Vietnamese youth.

Phase 2 will consist of a hybrid type 2 (where both implementation and clinical outcome measures are assessed), quasi-experimental, sequenced pre-post implementation design. The intervention takes a population-level approach to enhancing life skills and self-management skills that may be beneficial to all youth regardless of their mental health status. As this is a universal intervention, all students in grade 10 of participating secondary schools will be eligible to participate regardless of mental health and well-being status, as measured by standardized outcome measures. Control and intervention cohorts will be enrolled in each school in successive years. The control cohort will be recruited first and will be given the outcome assessments survey at baseline, 6 months, and 12 months marks. The control group will have access to the app after they have completed their final outcome assessment survey, but they will no longer provide outcome data and any in-app usage data (e.g. number and frequency of logins) which will be collected automatically by the app, will be excluded from the final analysis. The intervention cohort, recruited the year after the control cohort, will have full access to the app and will complete the same outcome measures at baseline, 6 and 12 months. Their app-usage data will be included in the final analysis.

The app-based intervention, co-designed with the V-YAC, aims to introduce life skills and self-management skills to promote general mental well-being and resilience among Vietnamese youth. With this app, youth users will have a fun and safe space to learn and practice six life skills areas (Problem-solving, Social Media and Well-being, Communication and Interpersonal Skills, Realistic Thinking, Coping with Emotions and Stress, and Goal Setting). Lessons (in the form of short texts) and activities (ex. multiple choice activities, blank worksheets, reflection questions) were adapted from evidence-based interventions developed in other contexts and were adapted in partnership with the V-YAC to ensure the skills and examples are culturally appropriate to the Vietnamese youth context. Youth users are free to explore the app at their own pace. Gamification features will also allow youth users to collect points in the app for completing each lesson, activity, or challenge (aimed to help encourage youth users to continue to practice skills after completing lessons). They then can use points to unlock and buy different accessories and backgrounds for their avatar (which is a gender neutral cartoon astronaut). Additionally, our app will include a mood check-in feature (where youth users can log and track their moods over time), guided breathing exercises, and a journaling feature.

Focus group discussions will be conducted with 6 - 8 participants at each school at the 12-month mark for each cohort to explore their experiences with the app, focusing on usability, appropriateness, and acceptability of app use. Semi-structured interviews with SHS, head teachers, and principals in each school will also be conducted to understand factors affecting implementation and potential scale-up of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in grade 10 of participating secondary schools
* Have access to a smartphone
* Provided informed assent to participate
* Parent of participant provided informed consent for their child to participate

Exclusion Criteria:

* Not in grade 10
* Not enrolled in participating secondary schools
* Not have access to a smartphone
* Not provided assent
* Parent did not provide consent

Ages: 15 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1800 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Warwick Edinburg Mental Wellbeing Scale (WEMWBS) | baseline, 6 months, 12 months
  The Warwick Edinburg Mental Wellbeing Scale (WEMWBS), a 14-item scale that uses positively worded statements to assess feeling and functioning aspects of mental well-being in the general population. Each item is rated on a 5-point Likert scale (1 = none of the time and 5 = all of the time). Higher sum scores indicate higher positive mental wellbeing.

SECONDARY OUTCOMES:
Positive Childhood Experience (PCE) | baseline, 6 months, 12 months
  The PCE score included 7 items adapted from the Child and Youth Resilience Measure. Each item is rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Higher sum scores indicate higher PCE.
Depression Anxiety and Stress Scale - Youth version (DASS -Y) | baseline, 6 months, 12 months
  The DASS-Y youth version of the DASS-21 is designed to measure general psychological distress and the negative emotional states of depression, anxiety and stress in youth (aged 7 - 18). Each of the 21 items is rated on a 4-point scale (1 = not true to 4 = very true). Higher sum scores indicate higher severity of symptoms.
Brief Inventory of Thriving (BIT) | baseline, 6 months, 12 months
  The BIT is a 10-item self-report questionnaire that measures positive functioning and well-being. Each item is rated on a 5-point scale (1 = strongly disagree to 5 = strongly agree). Higher sum scores indicate higher psychological well-being.
Connor-Davidson Resilience Scale - VN | baseline, 6 months, 12 months
  The Connor-Davidson Resilience Scale is a 10-item scale that measures resilience or the ability to bounce back from challenges. Each item is rated on a 5-point scale (0 = not true at all to 4 = true nearly all the time). Higher sum scores indicate higher levels of resilience.
Internet Addiction Test - Short version (S-IAT) | baseline, 6 months, 12 months
  The S-IAT consists of 12 questions that measures the frequency of problems related to internet overuse, focused on loss of control/time management and social problems. Each item is rated on a 5-point scale (1 = Never to 5 = Always). Higher sum scores indicate higher levels of internet addiction.
Educational Stress Scale for Adolescent (ESSA) | baseline, 6 months, 12 months
  The ESSA is a 16-item scale that measures level of academic-related stress. Each item is rated on a 5-point scale (1 = strongly disagree to 5 = strongly agree). Higher sum scores indicate greater stress
Alcohol & Substance Use, Bullying, Peer Influence, Punishment | baseline, 6 months, 12 months
  Items were adapted from the Vietnam Global Student Health Survey to measure use of the following items:
  * Alcohol & Substance Use: if the participant has ever used (and frequency) alcohol, cigarette, vape, nitric oxide, Vietnamese water pipe, shisha, and marijuana
  * Bullying: frequency and experiences of bullying and cyberbullying in the past 6 months
  * Peer Influence: presence of peer influence on alcohol and substance use
  * Punishment: frequency and method of discipline from parents and teachers in the past year
App Acceptability Scale | at 12 months
  5 items were adapted from the Acceptability of Health Apps among Adolescents to measure youth's acceptability of the current app. Each item is rated on a 5-point scale (1 = strongly disagree to 5 = strongly agree). Higher sum scores indicate higher levels of acceptability.
App usage data - implementation outcome | 6 months, 12 months
  Frequency of app log-in and duration of app engagement (how long are users using the app each time they open it Frequency and duration of feature engagement (how long are users interacting with each feature/lesson/activity)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Lam, MD, Principal Investigator — University of British Columbia; Jill Murphy, PhD, Principal Investigator — St. Francis Xavier University; Nguyen Vu, MD, Principal Investigator — Institute of Population Health and Development
Locations (1):
- Institute of Population, Health, and Development, Vietnam, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murphy JK, Nguyen VC, Linh DT, Xie H, Tran TH, Barbic SP, Chau LW, Samji H, Minas H, Nguyen MV, Obrzut A, O'Neil J, Michalak EE, Lam RW. Promoting mental well-being among secondary school students in Vietnam using the Y-MIND app: A protocol for a hybrid type 2, sequence pre-post, quasi-experimental study. PLoS One. 2025 Oct 7;20(10):e0332875. doi: 10.1371/journal.pone.0332875. eCollection 2025. PMID 41056276